CLINICAL TRIAL: NCT01028040
Title: Phase I, Single Centre, Open Label Study to Access The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous AZD3043 After A) a Single Ascending Bolus Dose and B) a Single Ascending Bolus Dose Followed by a Single Infusion Dose in Healthy Japanese Volunteers (Age Range 20-45 Years)
Brief Title: AZD Single Ascending Dose Study In Healthy Japanese Subjects
Acronym: JSAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D0510C00004
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Phase I; AZD3043; Japanese healthy volunteer
MeSH Terms: interventions — AZD-3043

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD3043 (Experimental)
  Interventions: Drug: AZD3043

INTERVENTIONS:
Drug: AZD3043 — Intravenous, single dose
Drug: AZD3043 — Infusion, single dose

SUMMARY:
This is a single centre, open label, non-randomised study to access the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD3043 following a single dose administration to Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male and females of non-childbearing potential aged ≥20 to ≤ 45 with suitable veins for cannulation or repeated venepuncture.
* Body weight 45-90 kg and Body mass index (BMI) ≥18.0 and ≤27.0 kg/m2
* Clinically normal physical findings including supine blood pressure, pulse rate, ECG, and laboratory assessments in relation to age, as judged by the Investigator.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically significant illness/infection or medical/surgical procedure or trauma, as judged by the Principal Investigator, within 4 weeks of the first administration of investigational product.
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis as judged by the Investigator

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD3043 following administration of SAD bolus (Part A) and SAD bolus followed by infusion (Part B). | From screening period to follow-up visit 42 days (Maximum)

SECONDARY OUTCOMES:
To characterize the PK of AZD3043 and its main metabolite (THRX-108893) & provisionally assess the dose-proportionality of the PK | Blood and urine sampling from pre-dose until follow-up visit, 10 days (approximately)
To evaluate the onset, level and recovery of/from sedation/anaesthesia. | Assessed on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ulrike Lorch, MFPM FRCA, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Research Site, London, United Kingdom